CLINICAL TRIAL: NCT05476679
Title: An Open Label Phase 2 Study to Evaluate the Effects of a Local Anesthetic, Anti-inflammatory Medications and Compression Garments on RZL-012-Induced Adverse Events
Brief Title: Evaluation the Effects of Various Treatments on RZL-012-Induced Adverse Events
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZL-012-SMF-SWMTG-001
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2022-07

CONDITIONS: Submental Fat
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RZL-012 50mg/ml (Experimental)
  Interventions: Drug: RZL-012; Drug: RZL-012+Lidacaine injection prior treatment; Drug: RZL-012+Medrol; Drug: RZL-012+Celecoxib+Zyrtec; Drug: RZL-012+facial and neck wrap

INTERVENTIONS:
Drug: RZL-012 — 50mg/ml drug formulation
Drug: RZL-012+Lidacaine injection prior treatment — 5ml lidocaine will be injected 10 minutes before RZL-012 treatment
Drug: RZL-012+Medrol — oral Medrol dose pack (8 mg (2 tablets) on Day 1 before treatment followed by 16 mg after treatment (as per Instructions for Use)). From Day 2, a daily tapering off by 4 mg until Day 6 will be administered per Rx Instructions for use
Drug: RZL-012+Celecoxib+Zyrtec — 200 mg Celecoxib BID and 10 mg Zyrtec BID on Days 1, 2, 3, 4, 5 and 6
Drug: RZL-012+facial and neck wrap — Universal Facial Band

SUMMARY:
This is a Phase 2, open-label, 2-stage, adaptive-design study in which subjects will be randomized into one of 5 treatment groups comprised of RZL-012 with or without additional study treatments:

DETAILED DESCRIPTION:
In the first stage of the study, 5 subjects will be randomized into each of the treatment groups. Study outcomes will be assessed up to one week thereafter to determine the need to modify additional study treatments. Subsequently up to 10 additional subjects will be randomized into each of the treatment groups for the second stage of the study.

For each subject, the study will consist of a screening period, baseline period in which subjects will receive a single treatment session of RZL-012 and a follow-up period. RZL-012 will be administered during a single treatment session via multiple injections into the submental area under the chin. Subjects will thereafter be monitored for safety and efficacy for at least 84 days.

Each subject will be treated with the same dose of RZL-012 :

• RZL-012 (concentration of injected solution 50 mg/mL RZL-012) of 7.5 mg/0.15 mL/injection point that results in a total dose/volume of 240±30mg mg/4.8±0.6 mL RZL-012, Each subject will receive additional study treatments in accordance with the treatment group to which the subject is randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female subject between the ages of 18 and 65 years, inclusive.
2. Has body mass index (BMI) between >22 kg/m2 and <40 kg/m2.
3. Has SMF bulge that is contiguous and fits to 32±4 injections sites according to a grid with 1 centimeter (cm) distance between injection points.
4. Has grade 3 to 4 of SMF as rated by both the C-CAT and S-CAT.
5. Has stable weight, with no fluctuation of >5 kg in the past 12 months.
6. If female, is not pregnant or breastfeeding based on the following:

   1. agree to the use of highly effective contraceptive methods for at least 2 weeks before baseline until 4 weeks after the last day of study drug and a negative serum pregnancy test (ß-hCG) at screening and negative urine pregnancy test at baseline; or
   2. is of nonchildbearing potential defined as clinically infertile as the result of surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy); or
   3. is confirmed postmenopausal status (defined as either having amenorrhea for ≥ 12 consecutive months without another cause and documented serum follicle-stimulating hormone (FSH) level > 40 mIU/mL or another documented medical condition (e.g., was born without a uterus)) NOTE: The following are considered highly effective contraceptive methods: hormonal oral contraceptives, injectables, and patches; intrauterine devices; double-barrier methods (synthetic condom, diaphragm, or cervical cap used with spermicidal foam, cream, or gel); and male partner sterilization.
7. If male (with or without vasectomy), agree to the use of highly effective contraceptive methods as listed above in criteria 7 as well as to use a barrier method, e.g. condom , from study check-in until 7 days after drug injection.
8. Is willing to avoid strenuous exercise for seven (7) days post treatment.
9. Is able to adhere to the visit schedule and protocol requirements and be available to complete the study.
10. Is willing and able to sign an Institutional Review Board (IRB) approved informed consent form (ICF) indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

1. Is unable to tolerate subcutaneous injections.
2. Has dysfunctional gallbladder activity (e.g., underwent cholecystectomy or cholecystitis).
3. Has any systemic disease including but not limited to gastritis or ulcers, renal dysfunction, hypertension, liver disease, glaucoma, diabetes and/or cardiovascular disease.
4. Has any contraindications to oral corticosteroids (prednisone), NSAIDs (e.g., Celecoxib) or non-sedative antihistamines (e.g. Zyrtec)
5. Has skin laxity (i.e., elastosis, skin crepiness, skin redundancy, skin draping, vertical and/or horizontal skin bands and folds, blunting of cervical mental angle, loss of opposition of skin to underlying neck structures due to skin laxity) that could obscure the evaluation and treatment of SMF.
6. Has any scars, unshaven hair, tattoos, facial hair or jewelry on or near the proposed treatment area.
7. Has presence of structures or confounding factors that may interfere with assessing SMF such as but not limited to enlarged submandibular salivary and/or parotid glands, micrognanthia, chin implant, soft tissue volume augmentation of chin and/or jawline, pronounced platysmal bands and deep necklace lines or presence of facial jowls that could obscure the evaluation of SMF.
8. Has a fat bulge under the chin that is too large to be adequately treated by 32±4 contiguous injections on a 1cm grid .
9. Has a fat bulge under the chin that is of an insufficient volume to allow 32±4 injections within a contiguous 1 cm grid.
10. Has significant history or current evidence of a medical, psychological or other disorder that, in the Investigator's opinion, would preclude enrollment in the study.
11. Has an active bacterial, fungal, or viral infection in the proposed treatment area.
12. Has a pre-existing skin condition in the submental region that, at the Investigator's discretion, may confound evaluation or analysis.
13. Has previously had treatments or surgery in the submentum, such as but not limited to, focused ultrasound, radiofrequency, cryolipolysis, liposuction, sodium deoxycholate, or neck lift.
14. Has pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia, or facial nerve palsy.
15. Has Dercum's Disease.
16. Has allergic reactions to injectables
17. Has allergic reactions to Zyrtec or Celecoxib.
18. Has any pre-existing medical condition other than increased SMF that, at the Investigator's discretion, may result in increased submental fullness, such as but not limited to, thyroid enlargement, goiter, cervical lymphadenopathy, etc.
19. Has a planned fat reduction procedure of any variety to the submental region for the duration of the study.
20. Has medication or a history of coagulopathy.
21. Has a history or family history of venous thrombotic disease.
22. Has been treated chronically at least three (3) months prior to study entry with systemic steroids or immunosuppressive drugs.
23. Has been treated chronically at least one (1) week prior to study entry with non-steroidal anti-inflammatory drugs (NSAIDs)
24. Has used anticoagulation therapies that may increase bleeding or bruising (i.e., aspirin, ibuprofen/Celecoxib, warfarin, vitamins, and herbal preparations) for seven (7) days prior to treatment.
25. .Has had treatment with botulinum toxin injections in the neck or chin area within nine (9) months prior to screening.
26. Current participation or participation within three (3) months prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luxurgery, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RZL-012+Lidacaine: RZL-012+Lidacaine injection prior treatment: 5ml lidocaine will be injected 10 minutes before RZL-012 treatment
Period: Overall Study
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidacaine | RZL-012+Medrol | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap
Started | 8 | 10 | 9 | 11 | 10
Completed | 8 | 10 | 9 | 9 | 10
Not Completed | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidacaine | RZL-012+Medrol | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap | Total
Number analyzed (Participants) | 8 | 10 | 9 | 11 | 10 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.9 (7.2) | 51.1 (8.6) | 49.8 (6.5) | 44 (9.5) | 36.8 (5.7) | 45.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 8 | 9 | 8 | 42
  Male | 0 | 1 | 1 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 9 | 11 | 10 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 1 | 2 | 4 | 11
  White | 5 | 7 | 8 | 8 | 6 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 9 | 11 | 10 | 48

OUTCOME MEASURES:

1. Primary Outcome: Safety - Adverse Events Follow up
Description: Number of subjects with severe swelling in each subgroup
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Groups:
- RZL-012+Methylprednisolone (Medrol): RZL-012+methylprednisolone (Medrol): oral Medrol dose pack (8 mg (2 tablets) on Day 1 before treatment followed by 16 mg after treatment (as per Instructions for Use)). From Day 2, a daily tapering off by 4 mg until Day 6 will be administered per Rx Instructions for use
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidacaine Injection Prior Treatment | RZL-012+Methylprednisolone (Medrol) | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap
Number analyzed (Participants) | 8 | 10 | 9 | 11 | 10
Participants | 1 | 2 | 3 | 0 | 0

2. Secondary Outcome: Efficacy -Reduction in Score According to Clinician Chin Assessment Tool (C-CAT)
Description: Number of subjects who has at least 1 grade improvement in C-CAT. The CAT is composed of 5 points where 0 represents no fat and 4 represent very noticeable bulge and fat that extends beyond the neck
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidacaine | RZL-012+Methylprednisolone (Medrol) | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap
Number analyzed (Participants) | 8 | 10 | 9 | 9 | 10
Participants | 6 | 10 | 9 | 8 | 9

3. Secondary Outcome: Efficacy - Number of Participants With 1 Grade Improvement According to the Subject Chin Assessment Tool (S-CAT)
Description: To determine the efficacy of RZL-012 vs. RZL-012 with additional treatments on Day 84 versus baseline using the Subject Chin Assessment Tool (S-CAT). The CAT is composed of 5 points where 0 represents no fat and 4 represent very noticeable bulge and fat that extends beyond the neck
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Groups:
- RZL-012+Lidocaine: RZL-012+Lidacaine injection prior treatment: 5ml lidocaine will be injected 10 minutes before RZL-012 treatment
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidocaine | RZL-012+Methylprednisolone (Medrol) | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap
Number analyzed (Participants) | 8 | 10 | 9 | 9 | 10
Participants | 4 | 3 | 6 | 6 | 5

4. Secondary Outcome: Efficacy - Percentage of Change From Baseline in Submental Fat Volume
Description: Percentage of change from baseline in submental fat volume , as measured with MRI in RZL-012 vs. RZL+other treatments treated subjects vs. placebo treated subjects on Day 84 following injection.
Time Frame: 84 days
Population: There were only 33/46 subjects that had an MRI scan.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidocaine | RZL-012+Methylprednisolone (Medrol) | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap
Number analyzed (Participants) | 6 | 6 | 7 | 8 | 6
percentage of change from baseline | -7.1 (6.0) | -15.4 (10.2) | -17.0 (12.9) | -10.8 (9.8) | -14.8 (7.6)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | RZL-012 50mg/ml | RZL-012+Lidacaine Injection Prior Treatment | RZL-012+Methylprednisolone (Medrol) | RZL-012+Celecoxib+Zyrtec | RZL-012+Facial and Neck Wrap
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/9 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/9 | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/8 | 10/10 | 9/9 | 11/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RZL-012 50mg/ml (N=8) | RZL-012+Lidacaine Injection Prior Treatment (N=10) | RZL-012+Methylprednisolone (Medrol) (N=9) | RZL-012+Celecoxib+Zyrtec (N=11) | RZL-012+Facial and Neck Wrap (N=10)
Hepatic mass, Liver function test increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RZL-012 50mg/ml (N=8) | RZL-012+Lidacaine Injection Prior Treatment (N=10) | RZL-012+Methylprednisolone (Medrol) (N=9) | RZL-012+Celecoxib+Zyrtec (N=11) | RZL-012+Facial and Neck Wrap (N=10)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 2 | 6 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 3 | 2 | 1 | 2
Injection site discomfort (General disorders) | 1 | 1 | 3 | 1 | 0
Injection site hemorrhage (General disorders) | 3 | 1 | 3 | 3 | 1
Injection site hypoesthesia (General disorders) | 1 | 4 | 2 | 2 | 2
Injection site induration (General disorders) | 0 | 1 | 0 | 1 | 0
Injection site oedema (General disorders) | 4 | 7 | 5 | 6 | 8
Injection site pain (General disorders) | 6 | 7 | 5 | 7 | 8
Injection site pruritus (General disorders) | 0 | 2 | 0 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Facial Paresis (General disorders) | 0 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT05476679/Prot_SAP_000.pdf